CLINICAL TRIAL: NCT01004380
Title: A Phase I Safety Study of Farletuzumab (MORAb-003), Carboplatin and Pegylated Liposomal Doxorubicin (PLD) in Subjects With Platinum-sensitive Ovarian Cancer
Brief Title: Safety Study of Farletuzumab, Carboplatin and Pegylated Liposomal Doxorubicin (PLD) to Treat Platinum-sensitive Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MORAb-003-005
Record Dates: First submitted 2009-10-20; First posted 2009-10-29 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Epithelial Ovarian Cancer; Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — farletuzumab; Carboplatin; 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Farletuzumab (Experimental): 2.5 mg/kg once weekly administered i.v. during the Combination treatment period and 7.5 mg/kg Q3W administered i.v. during the Maintenance period
  Interventions: Drug: Farletuzumab, Carboplatin, and PLD

INTERVENTIONS:
Drug: Farletuzumab, Carboplatin, and PLD — All subjects will receive approximately 6 cycles with carboplatin (AUC5-6) i.v. and PLD (30 mg/m2) i.v. on Day 1 of every 4-week Combination treatment cycle. In addition, subjects will also receive weekly farletuzumab at 2.5 mg/kg administered i.v. Following completion of the Combination treatment period (carboplatin/PLD/farletuzumab therapy),maintenance treatment with single agent farletuzumab will be administered once Q3W at 7.5 mg/kg until disease progression as defined by GCIG CA-125 (i.e., CA-125 is less than or equal to 2 × (ULN) documented on 2 occasions) or modified RECIST v.1.0 using CT or MRI.
  Other Names: Farletuzumab (MORAb-003); Carboplatin; PLD

SUMMARY:
The purpose of this study is to evaluate whether combination therapy with farletuzumab (MORAb-003), carboplatin, and pegylated liposomal doxorubicin (PLD) is safe.

DETAILED DESCRIPTION:
Farletuzumab (MORAb-003) is a monoclonal antibody that has the potential to be an effective agent against epithelial ovarian cancer (including primary fallopian tube and peritoneal adenocarcinoma) in combination with other drugs. Farletuzumab works by a different mechanism from other cancer therapeutics and has been shown to be well tolerated. This study allows the opportunity to determine if the combination therapy of farletuzumab, carboplatin, and PLD

1. is safe, or
2. to assess the potential drug-drug interaction, and
3. to prolong response to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epithelial ovarian cancer
* Must have measurable disease by CT or MRI scan
* Must have relapsed as defined by CA-125 or radiologically within 6 months or more of completion of first- or second-line platinum chemotherapy
* Must have been treated with surgery and be a candidate for repeat carboplatin therapy
* Must have a normal cardiac ejection fraction at baseline

Exclusion Criteria:

* Subjects who never responded to first- or second-line platinum-based chemotherapy or whose relapse occurs <6 months from the last platinum therapy
* Subjects who have received other therapy to treat their ovarian cancer since last relapse
* Known central nervous system tumor involvement
* Evidence of other active invasive malignancy
* Clinically significant heart disease
* Known allergic reaction to a prior monoclonal antibody therapy or have any documented HAHA
* Previous treatment with MORAb 003 (farletuzumab)
* Previous treatment with anthracyclines
* Clinical contraindications to use PLD

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the combination of farletuzumab, carboplatin, and PLD in subjects with platinum-sensitive ovarian cancer. | At all study visits.

SECONDARY OUTCOMES:
To assess the effect of farletuzumab in combination with carboplatin and PLD on best objective response rate, time to response, and duration of response by RECIST criteria. | Every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Weil, MD, Study Director — Morphotek
Locations (5):
- United States (5):
  - University of Alabama at Birmingham Medical Center, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland
  - Schwartz Gynecologic Oncology, Brightwaters, New York
  - Chattanooga GYN Oncology, Chattanooga, Tennessee
  - International Beneficence Clinical Research, LLC, Harlingen, Texas